CLINICAL TRIAL: NCT01281813
Title: Continued Access to Darunavir/Ritonavir (DRV/Rtv) in HIV-1 Infected Adults, Adolescents and Children Aged 3 Years and Above
Brief Title: TMC114IFD3001 - Study Providing Continued Access to Treatment With Darunavir (DRV)/Ritonavir(Rtv) in HIV1 Infected Adults, Adolescents and Children Aged 3 Years or Above and Coming From Previous Company Sponsored Studies With DRV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017230; TMC114IFD3001 (Other: Janssen Sciences Ireland UC); 2017-000285-30 (EudraCT Number); NCT03027297 (obsolete NCT alias)
Record Dates: First submitted 2010-12-30; First posted 2011-01-24 (Estimated); Results first posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: HIV-1 Infections
Keywords: TMC114IFD3001; TMC114; HIV; Darunavir; PREZISTA
MeSH Terms: interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Continued Treatment with DRV in Combination with rtv (Experimental): HIV-1 infected children participants (aged less than [<] 12 years) will continue to receive darunavir (DRV) 200 to 600 milligrams (mg) as oral suspension twice daily (BID) along with ritonavir (rtv) 32 to 100 mg as oral solution/suspension BID. HIV-1 infected adolescent participants (aged 12-17 years) will continue to receive DRV 200 to 600 mg as oral suspension BID along with rtv 32 to 100 mg as oral solution/suspension BID. Dosing for children and adolescent participants will be based on body weight (per parent study TMC114-TiDP29-C232). HIV-1 infected adult participants (aged greater than or equal to [>=] 18 years) will continue to receive DRV 800 mg (2 tablets of 400 mg) orally every day (qd) along with rtv 100 mg tablet (per parent study TMC114-C211) or DRV 600 mg tablet orally BID along with rtv 100 mg tablet (per parent study TMC114-C214 or TMC114-TiDP31-C229).
  Interventions: Drug: Darunavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Darunavir — Participants will receive darunavir (per parent study) as oral suspension.
Drug: Ritonavir — Participants will receive ritonavir (per parent study) as oral solution/suspension.

SUMMARY:
The primary objective of this trial is to continue the provision of darunavir/ low-dose ritonavir (DRV/rtv) to adult and pediatric patients who previously received DRV/rtv in the clinical trials TMC114-C211, TMC114-C214, TMC114-TiDP31-C229 or in the pediatric trial TMC114-TiDP29-C232 who continue to benefit from the use of darunavir in combination with low-dose ritonavir (DRV/rtv), in countries where DRV is not commercially available for the subject, is not reimbursed, or cannot be accessed through another source (e.g., access program, governmental program) and to provide DRV through this trial until the participants can switched to locally available DRV-based treatment regimens (that is commercially available and reimbursed, or accessible through another source [for example, access program or government program]) or to local standard of care, as appropriate.

DETAILED DESCRIPTION:
This is a continued access trial for adult and pediatric patients who have completed treatment with darunavir in combination with low-dose ritonavir (DRV/rtv) in the parent clinical trials TMC114-C211, TMC114-C214, TMC114-TiDP31-C229 or in the parent pediatric trial TMC114-TiDP29-C232 who continue to benefit from the use of DRV/rtv, and who live in a country where DRV is not accessible. At the baseline visit, inclusion and exclusion criteria will be checked to confirm eligibility. Once the eligibility criteria are met, patients will continue treatment as follows: HIV-1-infected patients participating in the TMC114-C211 trial and some HIV-1 infected patients from the pediatric trial TMC114-TiDP29-C232 will continue on the selected DRV/rtv once daily dosing regimen as administered in the original trial, or (for pediatric patients) on an adjusted dose if necessary due to a change in body weight. Some HIV-infected patients from the pediatric trial TMC114-TiDP29-C232 will continue on the selected twice daily DRV/rtv dosing regimen as administered in the original trial, or (for pediatric patients) on an adjusted dose if necessary due to a change in body weight. HIV-1-infected patients having participated in the TMC114-C214 or TMC114-TiDP31-C229 trial will continue on the DRV/rtv 600/100 mg twice daily dosing regimen as administered in the original trial. Visits and assessment are performed according to local standard of care, but desirable every 3 months for pediatric patients and not less frequently than every 6 months for adult patients. The interval between 2 consecutive visits should not exceed 6 months for pediatric patients. Adverse events (AEs) considered at least possibly related to DRV/rtv, AEs leading to discontinuation or treatment interruption, serious AEs (SAEs), and pregnancies (or all AEs if applicable per local regulation) will be recorded at each visit. Patients will be instructed to report any AEs to the investigator, who will report SAEs within 24 hours to the Sponsor. In addition to the assessments in the flowchart, the following assessments are recommended to be performed locally every 3 months or according to local, generally accepted standards of care: efficacy assessments (immunology and plasma viral load) and laboratory safety assessments (hematology and biochemistry, including pancreatic amylase [if available] or lipase and lipid analyses). Treatment will be continued until one of the following criteria is met (whichever occurs first): virologic failure; treatment-limiting toxicity; loss to follow-up; withdrawal of consent/assent by the patient; withdrawal of consent by the parent(s)/legal representative(s); pregnancy; termination of the trial by the sponsor; DRV based treatment regimen becomes commercially available for the patients and is reimbursed, or can be accessed through another source (for example, access program, government program) in the region the patient is living in or patients can be switched to local standard of care, as appropriate. A post-treatment follow-up contact is to be performed 4 weeks after the last dose of trial medication for patients with an ongoing adverse event, that discontinue the trial. This is consistent with the primary objective of the study to provide continued access to DRV/rtv for adult patients who previously received DR/rtv in the clinical trials sponsored by Tibotec Pharmaceuticals. This study is not set up to address any specific hypothesis. Depending on the previous trial the patients were in, they will continue to take either : DRV/rtv 800/100 mg once a day as 2 tablets of 400 mg DRV and 100 mg ritonavir; or DRV/rtv 600/100 mg twice a day as 1 tablet of 600 mg DRV and 100 mg ritonavir twice a day; DRV/rtv 375/100 mg twice a day as 1 tablet of 375 mg DRV and 100 mg ritonavir; DRV/rtv selected dose twice daily , or on an adjusted dose if necessary due to a change in body weight. For most of the patients, their next visit will be the final visit with data collection thereafter visits and assessments will be performed per local standard of care and documented in the patient's medical records only. Investigators will continue to report serious adverse events (SAEs) possibly related to DRV/rtv and pregnancies to the sponsor using regular reporting.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with DRV/rtv who have successfully completed the TMC114-C211, TMC114-C214, TMC114-TiDP31-C229 (parent) trial or the pediatric (parent) trial TMC114-TiDP29-C232 and in the opinion of the investigator continue to receive benefit from using DRV/rtv
* DRV is not commercially available for the patients, is not reimbursed, or cannot be accessed through another source (for example, access program, government program) in the region the patient is living in.
* Patients (where appropriate, depending on age) and the parent(s) or legal representative(s) have signed the Informed Consent/Assent Form voluntarily. Children will be informed about the program and asked to give assent (where appropriate, depending on age).

Exclusion Criteria:

* Any condition (including but not limited to alcohol and drug use) which, in the opinion of the investigator, could compromise the patient's safety or adherence to treatment with DRV/rtv
* Any active, clinically significant disease (such as pancreas or cardiac problems) or findings which could compromise the patient's safety during treatment with DRV/rtv
* Previously demonstrated clinically significant allergy or hypersensitivity to any of the excipients of the investigational medication (DRV) or ritonavir
* Pregnant or breastfeeding female patients

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2011-08-08 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (17):
- Rio de Janeiro, Brazil
- San José, Costa Rica
- Guatemala City, Guatemala
- Kuala Selangor, Malaysia
- Panama City, Panama
- South Africa (8):
  - Cape Town
  - Cyrildene Johannesburg Gauteng
  - Dundee
  - Durban
  - Johannesburg
  - Pretoria
  - Soweto
  - Westdene Johannesburg Gauteng
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
- Vinnitsa, Ukraine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had completed treatment with darunavir/ritonavir (DRV/rtv) in the adult clinical (parent) trials TMC114-C211 (NCT00258557), TMC114-C214 (NCT00110877), TMC114-TiDP31-C229 (NCT00524368) or in the pediatric (parent) trial TMC114-TiDP29-C232 (NCT01138605), who continued to benefit from the use of DRV/rtv, and who lived in a country where DRV was not accessible participated in this trial and continued treatment as per their respective parent study.
Pre-assignment Details: Adult participants who received either DRV/rtv 800/100 mg once daily or DRV/rtv 600/100 mg twice daily per parent study were included in single arm and combined analysis was performed as planned in protocol because the 2 doses were extensively evaluated in their respective parent studies (TMC114-C211,TMC114-C214 or TMC114-TiDP31-C229). Main purpose of this study was to provide continued access and not to compare the 2 doses (DRV/rtv 800/100 mg once daily or DRV/rtv 600/100 mg twice daily).
Groups:
- Continued Treatment With DRV in Combination With Rtv:Children Less Than (<) 12 Years: HIV-1 infected children participants with dose level carried over from the corresponding parent studies received darunavir (DRV) 200 to 600 milligrams (mg) as oral suspension twice daily (BID) along with ritonavir (rtv) 32 to 100 mg as oral solution/suspension BID based on their body weight (maximum exposure duration: up to 28 months).
- Continued Treatment With DRV in Combination With Rtv: Adolescents (12-17 Years): HIV-1 infected adolescent participants with dose level carried over from the corresponding parent studies received DRV 200 to 600 milligrams (mg) as oral suspension BID along with rtv 32 to 100 mg as oral solution/suspension BID based on their body weight (maximum exposure duration: up to 39 months).
- Continued Treatment With DRV in Combination With Rtv:Adults (Greater Than or Equal to [>=] 18 Years): HIV-1 infected adult participants with dose level carried over from the corresponding parent studies received DRV 800 mg (2 tablets of 400 mg) orally every day (qd) along with rtv 100 mg tablet (per parent study TMC114-C211) or DRV 600 mg tablet orally twice daily (BID) along with rtv 100 mg tablet (per parent study TMC114-C214 or TMC114-TiDP31-C229) (maximum exposure duration: up to 105 months).
Period: Overall Study
Arm/Group | Continued Treatment With DRV in Combination With Rtv:Children Less Than (<) 12 Years | Continued Treatment With DRV in Combination With Rtv: Adolescents (12-17 Years) | Continued Treatment With DRV in Combination With Rtv:Adults (Greater Than or Equal to [>=] 18 Years)
Started | 4 | 4 | 137
Completed | 0 | 0 | 0
Not Completed | 4 | 4 | 137
Not completed — Adverse Event | 0 | 0 | 10
Not completed — Lost to Follow-up | 0 | 0 | 31
Not completed — Withdrawal by Subject | 0 | 0 | 13
Not completed — Subject Non-Compliant | 0 | 0 | 6
Not completed — Subject Reached A Virologic Endpoint | 0 | 0 | 5
Not completed — Sponsor's Decision | 4 | 3 | 7
Not completed — Switched to Commercially Available Medication | 0 | 0 | 26
Not completed — Other | 0 | 1 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continued Treatment With DRV in Combination With Rtv:Children Less Than (<) 12 Years | Continued Treatment With DRV in Combination With Rtv: Adolescents (12-17 Years) | Continued Treatment With DRV in Combination With Rtv:Adults (Greater Than or Equal to [>=] 18 Years) | Total
Number analyzed (Participants) | 4 | 4 | 137 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 11 (0) | 13.8 (2.87) | 41.5 (8.6) | 39.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 82 | 85
  Male | 3 | 2 | 55 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 18 | 18
  Black or African American | 4 | 4 | 91 | 99
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 0 | 0 | 6 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
  Hispanic | 0 | 0 | 18 | 18
  Other | 0 | 0 | 4 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  BRAZIL | 0 | 1 | 0 | 1
  COSTA RICA | 0 | 0 | 7 | 7
  GUATEMALA | 0 | 0 | 4 | 4
  MALAYSIA | 0 | 0 | 3 | 3
  PANAMA | 0 | 0 | 8 | 8
  SOUTH AFRICA | 4 | 3 | 99 | 106
  THAILAND | 0 | 0 | 13 | 13
  UKRAINE | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Adverse events (AEs): any untoward medical occurrence (any unfavorable and unintended sign [including an abnormal laboratory finding], symptom, or disease) that occurred in a participant administered a pharmaceutical product and which did not necessarily have causal relationship with study treatment. Serious adverse events (SAEs): any untoward medical occurrence at any dose resulted: death; was life threatening; requires inpatient hospitalization/prolongation of existing hospitalization; resulted in persistent/significant disability/incapacity or congenital anomaly/birth defect. Adult participants who received either DRV/rtv 800/100 mg once daily or DRV/rtv 600/100 mg twice daily per parent study were included in single arm and combined analysis was performed as planned in protocol because the 2 doses were extensively evaluated in their respective parent studies. Main purpose of this study was to provide continued access and not to compare the 2 doses.
Time Frame: Up to 9 years 11 months
Population: Full Analysis Set (FAS) included all participants who had taken at least one dose of Darunavir (DRV), regardless of their compliance with the protocol and adherence to the dose regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Continued Treatment With DRV in Combination With Rtv:Children Less Than (<) 12 Years | Continued Treatment With DRV in Combination With Rtv: Adolescents (12-17 Years) | Continued Treatment With DRV in Combination With Rtv:Adults (Greater Than or Equal to [>=] 18 Years)
Number analyzed (Participants) | 4 | 4 | 137
Participants | 0 | 1 | 26

2. Primary Outcome: Number of Participants With Adverse Events Leading to Study Drug Discontinuation
Description: Adverse events (AEs) were defined as any untoward medical occurrence (any unfavorable and unintended sign [including an abnormal laboratory finding], symptom, or disease) that occurred in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adult participants who received either DRV/rtv 800/100 mg once daily or DRV/rtv 600/100 mg twice daily per parent study were included in single arm and combined analysis was performed as planned in protocol because the 2 doses were extensively evaluated in their respective parent studies. Main purpose of this study was to provide continued access and not to compare the 2 doses.
Time Frame: Up to 9 years 11 months
Population: FAS included all participants who had taken at least one dose of DRV, regardless of their compliance with the protocol and adherence to the dose regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Continued Treatment With DRV in Combination With Rtv:Children Less Than (<) 12 Years | Continued Treatment With DRV in Combination With Rtv: Adolescents (12-17 Years) | Continued Treatment With DRV in Combination With Rtv:Adults (Greater Than or Equal to [>=] 18 Years)
Number analyzed (Participants) | 4 | 4 | 137
Participants | 0 | 0 | 9

3. Primary Outcome: Number of Participants With Adverse Events Possibly Related to Darunavir/Ritonavir (DRV/Rtv) Treatment
Description: Number of participants with adverse events possibly related to DRV/rtv treatment were reported. Adult participants who received either DRV/rtv 800/100 mg once daily or DRV/rtv 600/100 mg twice daily per parent study were included in single arm and combined analysis was performed as planned in protocol because the 2 doses were extensively evaluated in their respective parent studies. Main purpose of this study was to provide continued access and not to compare the 2 doses.
Time Frame: Up to 9 years 11 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Continued Treatment With DRV in Combination With Rtv:Children Less Than (<) 12 Years | Continued Treatment With DRV in Combination With Rtv: Adolescents (12-17 Years) | Continued Treatment With DRV in Combination With Rtv:Adults (Greater Than or Equal to [>=] 18 Years)
Number analyzed (Participants) | 4 | 4 | 137
Participants | 0 | 0 | 4

ADVERSE EVENTS:
Time Frame: Up to 9 years 11 months
Description: Full Analysis Set: participants had at least 1 dose DRV, regardless of protocol compliance and dose regimen adherence. Adult participants who received either DRV/rtv 800/100 mg once daily or DRV/rtv 600/100 mg twice daily per parent study included in single arm and combined analysis was performed as planned in protocol since the 2 doses were extensively evaluated in their respective parent studies. Main purpose of this study was to provide continued access and not to compare the 2 doses.
Arm/Group | Continued Treatment With DRV in Combination With Rtv:Children Less Than (<) 12 Years | Continued Treatment With DRV in Combination With Rtv: Adolescents (12-17 Years) | Continued Treatment With DRV in Combination With Rtv:Adults (Greater Than or Equal to [>=] 18 Years)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 3/137
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4 | 26/137
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 4/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continued Treatment With DRV in Combination With Rtv:Children Less Than (<) 12 Years (N=4) | Continued Treatment With DRV in Combination With Rtv: Adolescents (12-17 Years) (N=4) | Continued Treatment With DRV in Combination With Rtv:Adults (Greater Than or Equal to [>=] 18 Years) (N=137)
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1
Deafness Unilateral (Ear and labyrinth disorders) | 0 | 0 | 1
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Bone Tuberculosis (Infections and infestations) | 0 | 0 | 1
Breast Abscess (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Groin Abscess (Infections and infestations) | 0 | 0 | 1
Infected Cyst (Infections and infestations) | 0 | 0 | 1
Malaria (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2
Pulmonary Tuberculosis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 2
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foetal Exposure During Pregnancy (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Maternal Exposure During Breast Feeding (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Abortion Threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Foetal Death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Premature Baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Premature Labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Acute Psychosis (Psychiatric disorders) | 0 | 0 | 1
Intentional Self-Injury (Psychiatric disorders) | 0 | 1 | 0
Major Depression (Psychiatric disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 0 | 3
Immature Respiratory System (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Continued Treatment With DRV in Combination With Rtv:Children Less Than (<) 12 Years (N=4) | Continued Treatment With DRV in Combination With Rtv: Adolescents (12-17 Years) (N=4) | Continued Treatment With DRV in Combination With Rtv:Adults (Greater Than or Equal to [>=] 18 Years) (N=137)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT01281813/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT01281813/SAP_001.pdf